CLINICAL TRIAL: NCT03419104
Title: Use of Preoperative Exercise Test as Predictor for Postoperative Intensive Care Unit Need in Patients Undergoing Bariatric Surgery
Brief Title: Preoperative Exercise Test and Postoperative Intensive Care Unit Need in Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, Prof.Dr, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IstanbulU ctf
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Morbid Obesity; Weaning Failure
Keywords: bariatric surgery; extubation
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative walk test (Experimental): Patients undergoing bariatric surgery who will complete a preoperative 60 meters 60 seconds walk test.
  Interventions: Diagnostic Test: preoperative walk test

INTERVENTIONS:
Diagnostic Test: preoperative walk test — Patients undergoing bariatric surgery who will complete a preoperative 60 meters 60 seconds walk test.

SUMMARY:
The aim of our study is to evaluate the efficacy of "60 meters 60 seconds exercise test" (a test designed by the study group) done preoperatively as a predictor test for postoperative intensive care unit need and extubation success in patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

patients between 18-60 years old patients with BMI > 40 patients undergoing Laparoscopic Sleeve Gastrectomy

Exclusion Criteria:

patients with Chronic obstructive pulmonary disease (COPD) or Asthma, patients with uncompensated heart failure Patients Who have orthopedic problems that effects the exercise test (such as gonarthrosis)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
extubation | one hour postoperative
  Number of participants with successful extubation and patients who does not need mechanical ventilation support

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gupta PK, Gupta H, Kaushik M, Fang X, Miller WJ, Morrow LE, Armour-Forse R. Predictors of pulmonary complications after bariatric surgery. Surg Obes Relat Dis. 2012 Sep-Oct;8(5):574-81. doi: 10.1016/j.soard.2011.04.227. Epub 2011 May 13. PMID 21719358